CLINICAL TRIAL: NCT06458920
Title: Social Facilitation of Emotion Regulation in Adolescence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jennifer Silvers, PhD, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21-000929; R21HD108751 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation | interventions — Social Control, Formal

STUDY DESIGN:
Intervention Model Description: During one MRI scan, participants will spend part of the time regulating emotion on their own and part of the time regulating emotion with the help of a friend
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Social regulation (Experimental): Participants will regulate emotion with the help of a friend
  Interventions: Behavioral: Social regulation
- Cognitive regulation (Experimental): Participants will regulate emotion on their own
  Interventions: Behavioral: Cognitive regulation

INTERVENTIONS:
Behavioral: Social regulation — Participants will regulate emotion with the help of a friend
  Arms: Social regulation
Behavioral: Cognitive regulation — Participants will regulate emotion on their own
  Arms: Cognitive regulation

SUMMARY:
The goal of this project is to test whether regulating emotions with help from a friend is more effective and long-lasting in adolescents than regulating alone, and to characterize age-related differences in the neural mechanisms supporting social versus cognitive emotion regulation. Participants will complete a psychology experiment while undergoing fMRI scanning.

DETAILED DESCRIPTION:
Participants will complete a novel paradigm during functional magnetic resonance imaging (fMRI) to examine whether adolescents (N = 50) and adults (N = 50) are more effective at down-regulating negative affect when a friend provides them with reinterpretations of negative stimuli (i.e. social reappraisal), as compared to when they reinterpret stimuli alone (i.e., cognitive reappraisal). Specifically, participants will look at pictures of upsetting events while undergoing fMRI scanning. For some pictures, they will be instructed to just look at the image. For other pictures, they will be told to listen to their friend's voice as their friend helps them to regulate their emotions. For other pictures, they will be told to regulate their emotions on their own. The primary comparison of interest is how participants regulate emotion on their own versus when their friend helps them.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent participants must be 13-15 year of age
* Adult participants must be 20-25 years of age
* Proficient in English

Exclusion Criteria:

* Auditory, visual or cognitive impairment
* Any health conditions that are contraindicated for MRI

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Negative affect | 1 day
  Participant's self-reported negative affect on 1-4 scale (1=not bad at all, 4=very bad) during experiment

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data including age, gender and negative affect
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 12 months from study completion
Access Criteria: Deidentified data will be posted on Open Science Framework